CLINICAL TRIAL: NCT01468987
Title: The Impact of LY2605541 Versus Insulin Glargine for Patients With Type 2 Diabetes Mellitus Advanced to Multiple Injection Bolus Insulin With Insulin Lispro: a Double-Blind, Randomized, 26-week Study - The IMAGINE 4 Study
Brief Title: A Study in Participants With Type 2 Diabetes Mellitus
Acronym: IMAGINE 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12145; I2R-MC-BIAM (Other: Eli Lilly and Company); 2011-001254-29 (EudraCT Number)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2605541; basal insulin peglispro; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Glargine + Insulin Lispro (Active Comparator): Participant-specific dose of Insulin Glargine will be administered subcutaneously (SC) once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro will be administered SC for preprandial (pre-meal) and supplemental doses for 26 weeks.
  Interventions: Drug: Insulin Glargine; Drug: Insulin Lispro
- LY2605541 + Insulin Lispro (Experimental): Participant-specific dose of LY2605541 will be administered SC once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro will be administered SC for preprandial and supplemental doses for 26 weeks.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY2605541
  Other Names: Insulin Peglispro
  Arms: LY2605541 + Insulin Lispro
Drug: Insulin Glargine
  Arms: Insulin Glargine + Insulin Lispro
Drug: Insulin Lispro
  Other Names: Humalog

SUMMARY:
The purpose of this study is:

* To compare blood glucose (blood sugar) control on LY2605541 with insulin glargine after 26 weeks of treatment.
* To compare the rate of night time hypoglycemia (low blood glucose) on LY2605541 with insulin glargine during 26 weeks of treatment.
* To compare the number of participants on LY2605541 reaching blood glucose targets without hypoglycemia episodes at night to those taking insulin glargine after 26 weeks of treatment.
* To compare the rate of hypoglycemia over a 24-hour period on LY2605541 with insulin glargine during 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria

* Have type 2 diabetes mellitus based on the World Health Organization (WHO) classification
* Had diabetes ≥1 year
* Have a hemoglobin A1c (HbA1c) value ≥7.0% and <12.0% at screening
* Have a body mass index (BMI) ≤45.0 kilograms per square meter (kg/m^2)
* Participants on any glucose lowering regimen that contains at least 1 daily insulin injection
* This inclusion criterion applies ONLY to women of childbearing potential

  * Are not breastfeeding
  * Test negative for pregnancy at screening and randomization
  * Do not intend to become pregnant during the study
  * Have practiced a reliable method of birth control for at least 6 weeks prior to screening
  * Agree to continue to use a reliable method of birth control during the study, as determined by the investigator (and for 2 weeks following the last dose of study drug)
* Have access to a method of communication with the site
* Have refrigeration in the home
* Capable of, and willing to do the following: adhere to a multiple daily injection regimen, inject insulin with a covered vial and syringe and prefilled pen, attend some appointments in the fasting state, and perform self blood glucose monitoring and record keeping as required by this protocol, as determined by the investigator. Caregiver may be responsible for all of the above
* Have given written informed consent to participate in this study in accordance with local regulations

Exclusion Criteria

* Continuous subcutaneous insulin infusion therapy prior to screening
* Are using twice daily insulin glargine prior to screening
* Excessive insulin resistance defined as having received a daily dose of insulin ≥2.0 units per kilogram (units/kg) at the time of pre-randomization
* Glucagon-like peptide-1 (GLP-1) receptor agonist (eg, exenatide, exenatide once weekly, or liraglutide), thiazolidinedione (rosiglitazone, pioglitazone), or pramlintide, used concurrently or within 90 days prior to screening
* Are using niacin preparations as a lipid-lowering medication and/or bile acid sequestrants within 90 days prior to screening; or, are using lipid-lowering medication at a dose that has not been stable for ≥90 days prior to screening
* Have fasting hypertriglyceridemia (defined as >4.5 millimoles per liter [mmol/L], >400 milligrams per deciliter [mg/dL]) at screening
* Are currently taking, or have taken within the 90 days preceding screening, prescription or over-the-counter medications for weight loss
* Have had any episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within 6 months prior to entry into the study
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control within the 6 months prior to screening
* Have had 1 or more episodes of ketoacidosis or hyperosmolar state/coma requiring hospitalization within 6 months prior to screening
* Have cardiac disease with functional status that is New York Heart Association Class III or IV (per New York Heart Association Cardiac Disease Classification)
* Are currently receiving renal dialysis or have a serum creatinine ≥2.0 mg/dL, except for participants taking metformin who will be required to follow local labeling restrictions regarding metformin use and serum creatinine
* Have obvious clinical signs or symptoms of liver disease (excluding non-alcoholic fatty liver disease [NAFLD], acute or chronic hepatitis, non-alcoholic steatohepatitis [NASH], or elevated liver enzyme measurements as indicated below:

  * total bilirubin ≥2X the upper limit of normal (ULN) as defined by the central laboratory, or
  * alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) >2.5X ULN as defined by the central laboratory, or
  * aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) >2.5X ULN as defined by the central laboratory
* Have active or untreated malignancy, have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years, or are at increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
* Have known or develop hypersensitivity or allergy to any of the study insulins or their excipients
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the HbA1c measurement
* Receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, and inhaled preparations) or have received such therapy within 8 weeks immediately before screening with the exception of replacement therapy for adrenal insufficiency
* Diagnosed clinically significant diabetic autonomic neuropathy, in the opinion of the investigator
* Have had an organ transplant
* Have any other condition (including known drug or alcohol abuse or psychiatric disorder including eating disorder) that precludes the participant from following and completing the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1369 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (155):
- United States (48):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chino, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longmont, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Haven, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagan, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jefferson City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mentor, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
- Australia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camperdown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daw Park, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Ringwood, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geelong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremantle, Western Australia
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aparecida de Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasília
- Croatia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Čakovec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rijeka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slavonski Brod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varaždin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hranice I-Mesto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krnov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esbjerg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hillerød
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burghausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eisenach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falkensee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuwied
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nikaias - Piraeus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- Israel (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beersheba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nahariya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Safed
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pavia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Querétaro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Netherlands (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dordrecht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heerlen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoogeveen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Lomas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yabucoa
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Satu Mare
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dolný Kubín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ľubochňa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rožňava
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yong Kung City
- Turkey (Türkiye) (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Diyarbakır
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kütahya
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlesbrough, Cleveland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester, Leicestershire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541 + Insulin Lispro: Includes participants that were randomized to receive LY2605541 plus Insulin Lispro.
  Participant-specific dose of LY2605541 was administered subcutaneously (SC) once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro was administered SC for preprandial (pre-meal) and supplemental doses for 26 weeks.
- Insulin Glargine + Insulin Lispro: Includes participants that were randomized to receive Insulin Glargine plus Insulin Lispro.
  Participant-specific dose of Insulin Glargine was administered SC once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro was administered SC for preprandial and supplemental doses for 26 weeks.
Period: Overall Study
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Started | 691 | 678
Received at Least 1 Dose of Study Drug | 691 | 677
Completed | 620 | 618
Not Completed | 71 | 60
Not completed — Adverse Event | 12 | 9
Not completed — Death | 4 | 1
Not completed — Lost to Follow-up | 10 | 5
Not completed — Protocol Violation | 8 | 2
Not completed — Withdrawal by Subject | 28 | 28
Not completed — Physician Decision | 8 | 15
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- LY2605541 + Insulin Lispro: Participant-specific dose of LY2605541 was administered SC once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro was administered SC for preprandial and supplemental doses for 26 weeks.
- Insulin Glargine + Insulin Lispro: Participant-specific dose of Insulin Glargine was administered SC once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro was administered SC for preprandial and supplemental doses for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro | Total
Number analyzed (Participants) | 691 | 678 | 1369
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.43 (9.21) | 57.77 (9.17) | 57.6 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 274 | 589
  Male | 376 | 404 | 780
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 78 | 152
  Not Hispanic or Latino | 452 | 427 | 879
  Unknown or Not Reported | 165 | 173 | 338
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 25 | 30 | 55
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 42 | 50 | 92
  White | 615 | 585 | 1200
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 276 | 270 | 546
  Taiwan | 7 | 8 | 15
  Slovakia | 25 | 17 | 42
  Greece | 12 | 11 | 23
  Spain | 30 | 35 | 65
  Lithuania | 4 | 2 | 6
  Turkey | 4 | 7 | 11
  Austria | 9 | 6 | 15
  Russia | 19 | 20 | 39
  Israel | 20 | 20 | 40
  United Kingdom | 5 | 3 | 8
  Italy | 16 | 16 | 32
  Czechia | 23 | 22 | 45
  Hungary | 36 | 36 | 72
  Mexico | 13 | 12 | 25
  Puerto Rico | 20 | 26 | 46
  Poland | 20 | 20 | 40
  Brazil | 11 | 13 | 24
  Romania | 34 | 31 | 65
  Croatia | 5 | 2 | 7
  Denmark | 9 | 3 | 12
  Australia | 26 | 25 | 51
  Netherlands | 7 | 8 | 15
  Germany | 50 | 54 | 104
  Japan | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at 26 Weeks
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2 to 3 month timeframe. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for stratification factors (country, low-density lipoprotein cholesterol [LDL-C, <100 milligrams per deciliter (mg/dL) and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), visit, treatment, visit-by-treatment interaction, and baseline HbA1c.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 684 | 672
percentage of HbA1c | -1.66 (0.04) | -1.45 (0.04)

2. Secondary Outcome: Total Hypoglycemia Rates (Adjusted for 30 Days)
Description: Hypoglycemic episodes are defined as events which are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 millimoles per liter [mmol/L]). Group mean rates of total hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline total hypoglycemia rate, with log [exposure in days/30] as an offset variable). Group Mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable data at both baseline and post-baseline.
Measure: Mean (Standard Error); unit: episodes/participant/30 days
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 689 | 676
episodes/participant/30 days | 5.97 (0.20) | 5.42 (0.19)

3. Secondary Outcome: Percentage of Participants With Total Hypoglycemia Episodes
Description: Hypoglycemic episodes are defined as events which are associated with reported signs and symptoms of hypoglycemia and/or documented BG concentrations of ≤70 mg/dL (3.9 mmol/L). The percentage of participants was calculated by dividing the number of participants with hypoglycemic episodes by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline through 26 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 689 | 676
percentage of participants | 95.2 | 96.6

4. Secondary Outcome: Nocturnal Hypoglycemia Rates (Adjusted for 30 Days)
Description: Hypoglycemic episodes are defined as events which are associated with reported signs and symptoms of hypoglycemia and/or a documented BG concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. Group mean rates of nocturnal hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline nocturnal hypoglycemia rate, with log [exposure in days/30] as an offset variable). Group Mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: events/participant/30 days
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 689 | 676
events/participant/30 days | 0.51 (0.03) | 0.92 (0.05)

5. Secondary Outcome: Percentage of Participants With Nocturnal Hypoglycemia Episodes
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia and/or a BG concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. The percentage of participants was calculated by dividing the number of participants with nocturnal hypoglycemic episodes by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline through 26 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Insulin Glargine + Insulin Lispro: Participant-specific dose of Insulin Glargine were administered SC once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro were administered SC for preprandial and supplemental doses for 26 weeks.
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 689 | 676
percentage of participants | 59.5 | 74.0

6. Secondary Outcome: Body Weight Change From Baseline to 26 Weeks
Description: LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), treatment, visit, treatment-by-visit interaction, and baseline body weight as fixed effects, and participant as a random effect.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable body weight data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 682 | 671
kilograms (kg) | 1.25 (0.16) | 2.21 (0.16)

7. Secondary Outcome: Self-Monitored Blood Glucose (SMBG) 9-point Profiles at 26 Weeks
Description: 9-point SMBG profiles were obtained over 2 nonconsecutive days within the week prior to Weeks 0, 4, 12, and 26. SMBG measurements were taken at 9 time points: pre-morning meal, 2 hours post-morning meal, pre-midday meal, 2 hours post-midday meal, pre-evening meal, 2 hours post-evening meal, bedtime, at approximately 0300 hours, and the subsequent morning prior to the morning meal. LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), visit, treatment, visit-by-treatment interaction, and baseline BG values.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 639 | 619
mg/dL
  Pre-morning meal | 137.31 (1.63) | 133.81 (1.66)
  2 hours post-morning meal: number analyzed (Participants) | 545 | 538
  2 hours post-morning meal | 162.77 (2.59) | 156.41 (2.64)
  Pre-midday meal: number analyzed (Participants) | 606 | 584
  Pre-midday meal | 130.02 (1.97) | 133.63 (2.02)
  2 hours post-midday meal: number analyzed (Participants) | 548 | 550
  2 hours post-midday meal | 145.55 (2.67) | 156.17 (2.72)
  Pre-evening meal: number analyzed (Participants) | 611 | 595
  Pre-evening meal | 142.65 (2.09) | 149.19 (2.14)
  2 hours post-evening meal: number analyzed (Participants) | 552 | 536
  2 hours post-evening meal | 156.56 (2.72) | 166.59 (2.85)
  Bedtime: number analyzed (Participants) | 587 | 557
  Bedtime | 160.15 (2.60) | 163.62 (2.70)
  0300 hours: number analyzed (Participants) | 516 | 487
  0300 hours | 143.90 (2.54) | 140.19 (2.59)
  Pre-morning meal next day: number analyzed (Participants) | 605 | 588
  Pre-morning meal next day | 135.09 (1.77) | 132.07 (1.81)

8. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and ≤6.5% at 26 Weeks
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: up to 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 684 | 672
percentage of participants
  HbA1c ≤6.5% | 44.4 | 32.6
  HbA1c <7.0% | 63.3 | 53.3

9. Secondary Outcome: Percentage of Participants With HbA1c <7.0% Without Nocturnal Hypoglycemia at 26 Weeks
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia and/or a documented blood glucose concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking and between the time points of 10:00 PM and 10:00 AM. The percentage of participants was calculated by dividing the number of participants with HbA1c <7.0% without nocturnal hypoglycemia by the total number of participants analyzed, multiplied by 100.
Time Frame: up to 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data. Missing endpoints were imputed with the LOCF method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Groups:
- LY2605541 + Insulin Lispro: Participant-specific dose of LY2605541 was administered SC once daily at bedtime for 26 weeks.
  Participant-specific dose of Insulin Lispro were administered SC for preprandial and supplemental doses for 26 weeks.
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 684 | 672
percentage of participants | 23.7 | 12.2

10. Secondary Outcome: Basal, Bolus, and Total Insulin Dose by Weight at 26 Weeks
Description: Basal insulin dose, short-acting bolus insulin dose (each meal and overall), and total insulin dose were calculated based on the dose during the last 7 days prior to the post-treatment visit or last 3 days prior to the randomization visit. LS means were calculated using a constrained Longitudinal Data Analysis (cLDA) model adjusting for indicator variables of each treatment group at each post-baseline visit and stratification variables (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and baseline number of insulin injections [1, 2, or ≥3]).
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units/kg/day
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 615 | 613
units/kg/day
  Basal Insulin: number analyzed (Participants) | 612 | 606
  Basal Insulin | 0.68 (0.01) | 0.60 (0.01)
  Bolus Insulin: number analyzed (Participants) | 591 | 591
  Bolus Insulin | 0.61 (0.02) | 0.63 (0.02)
  Total Insulin | 1.27 (0.02) | 1.21 (0.02)

11. Secondary Outcome: Fasting Serum Glucose (FSG) From Laboratory at 26 Weeks
Description: LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), treatment, visit, treatment-by-visit interaction, and baseline FSG.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FSG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 683 | 672
mg/dL | 125.33 (1.93) | 132.02 (1.94)

12. Secondary Outcome: Fasting Blood Glucose (FBG) (by SMBG) Intra-participant Variability at 26 Weeks
Description: FBG was measured by self-monitored blood glucose (SMBG). Between-day glucose variability is measured by the standard deviation of FBG. LS means were calculated using MMRM adjusting for the stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), treatment, visit, treatment-by-visit interaction, and baseline FBG variability.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 674 | 652
mg/dL | 28.67 (0.79) | 33.54 (0.80)

13. Secondary Outcome: 0300-hour Blood Glucose to FBG Excursion at 26 Weeks
Description: Results of a 0300-hour to pre-morning meal (FBG) excursion are presented (only SMBG profiles with both 0300 hours and the next day pre-morning measurements are included for the calculation of such excursion). LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), treatment, visit, treatment-by-visit interaction, and baseline excursion.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 470 | 450
mg/dL | -11.95 (2.34) | -15.16 (2.37)

14. Secondary Outcome: HbA1c at 26 Weeks
Description: HbA1c is a test that measures a participant's average blood glucose level over the past 2 to 3 months. LS means were calculated using MMRM adjusting for stratification factors (country, LDL-C [<100 mg/dL and ≥100 mg/dL], and number of insulin injections at baseline [1, 2, or ≥3]), treatment, visit, treatment, visit-by-treatment interaction, and baseline HbA1c.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 684 | 672
percentage of HbA1c | 6.76 (0.04) | 6.97 (0.04)

15. Secondary Outcome: Lipid Profile at 26 Weeks
Description: Concentrations of cholesterol, high-density lipoprotein cholesterol (HDL-C), LDL-C, and triglycerides are summarized. LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL and ≥100 mg/dL], except for the LDL-C outcome variable], number of insulin injections at baseline [1, 2, or ≥3]), visit, treatment, visit-by-treatment interaction, and baseline value of corresponding lipid outcome variable.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable lipid data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 684 | 674
mg/dL
  Cholesterol: number analyzed (Participants) | 613 | 609
  Cholesterol | 177.17 (1.13) | 174.79 (1.14)
  HDL-C: number analyzed (Participants) | 611 | 603
  HDL-C | 46.44 (0.27) | 47.71 (0.27)
  LDL-C: number analyzed (Participants) | 609 | 603
  LDL-C | 97.87 (0.99) | 98.89 (0.99)
  Triglycerides: number analyzed (Participants) | 614 | 609
  Triglycerides | 168.79 (2.85) | 141.78 (2.86)

16. Secondary Outcome: Number of Participants With Change in Anti-LY2605541 Antibodies From Baseline to 26 Weeks
Description: The number of participants with a treatment-emergent anti-LY2605541 antibody response (TEAR) is summarized. TEAR is defined as change from baseline to post-baseline in the anti-LY2605541 antibody level either from undetectable to detectable, or from detectable to the value with at least 130% relative increase from baseline.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable anti-LY2605541 antibody data at baseline and post-baseline.
Measure: Number; unit: participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 682 | 672
participants | 152 | 161

17. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) at 26 Weeks
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where higher scores indicate better treatment satisfaction. LS means were calculated using an analysis of covariance (ANCOVA) model with treatment and stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, and baseline number of insulin injections [1, 2, or ≥3]) as fixed effects and baseline value of the ITSQ scores as a covariate.
Time Frame: up to 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable ITSQ data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 631 | 637
units on a scale | 77.01 (0.55) | 77.29 (0.54)

18. Secondary Outcome: Low Blood Sugar Survey (LBSS) at 26 Weeks
Description: LBSS (also referenced as Hypoglycemia Fear Survey - II [HFS-II]) is a 33-item questionnaire that measures 1) behaviors to avoid hypoglycemia and its negative consequences (15 items) and 2) worries about hypoglycemia and its negative consequences (18 items). Responses are made on a 5-point Likert scale where 0 = Never and 4 = Always. Total score is the sum of all items (range 0-132). Higher total scores reflect greater fear of hypoglycemia. LS means were calculated using MMRM including stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, baseline number of insulin injections [1, 2, or ≥3]), visit, treatment, visit-by-treatment interaction, and baseline LBSS score.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable LBSS data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 682 | 671
units on a scale | 21.44 (0.56) | 21.67 (0.56)

19. Secondary Outcome: EuroQoL-5D (EQ-5D) at 26 Weeks
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a three level scale of 1-3 (no problem, some problems, and extreme problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United States population-based algorithm. Scores range from -0.11 to 1.0, where a score of 1.0 indicates perfect health. LS means were calculated using ANCOVA adjusting for treatment, stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, and baseline number of insulin injections [1, 2, or ≥ 3]), and baseline EQ-5D score.
Time Frame: up to 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable EQ-5D data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 636 | 644
units on a scale | 0.86 (0.00) | 0.85 (0.00)

20. Secondary Outcome: Rapid Assessment of Physical Activity (RAPA) at 26 Weeks
Description: The RAPA questionnaire assesses the level and intensity of physical activity of adult participants. It contains 2 subscales: RAPA 1 (Aerobic) and RAPA 2 (Strength and Flexibility). RAPA 1 contains 7 questions regarding the participant's amount and intensity of physical activity, allowing each participant's aerobic activity level to be categorized as sedentary, underactive, light activities, light activity, regular underactive, or active. RAPA 2 contains 2 questions regarding participants' physical activities that increase strength and improve flexibility. Each participant's strength and flexibility activity level is then categorized as neither strength nor flexibility activity, either strength or flexibility activity (not both), both strength and flexibility activity. The percentage of participants in each RAPA 1/2 category is presented and was calculated by dividing the number of participants in each RAPA 1/2 category by the total number of participants analyzed, multiplied by 100.
Time Frame: up to 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable RAPA data. Missing endpoints were imputed with the LOCF method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Number analyzed (Participants) | 331 | 346
percentage of participants
  RAPA 1, Sedentary: number analyzed (Participants) | 324 | 339
  RAPA 1, Sedentary | 2.2 | 2.4
  RAPA 1, Underactive: number analyzed (Participants) | 324 | 339
  RAPA 1, Underactive | 4.6 | 6.2
  RAPA 1, Light activity: number analyzed (Participants) | 324 | 339
  RAPA 1, Light activity | 21.9 | 18.0
  RAPA 1, Regular underactive: number analyzed (Participants) | 324 | 339
  RAPA 1, Regular underactive | 32.7 | 27.1
  RAPA 1, Active: number analyzed (Participants) | 324 | 339
  RAPA 1, Active | 38.6 | 46.3
  RAPA 2, Neither strength/flexibility | 58.3 | 53.8
  RAPA 2, Either strength/flexibility | 28.1 | 30.6
  RAPA 2, Both strength/flexibility | 13.6 | 15.6

ADVERSE EVENTS:
Groups:
- LY2605541 + Insulin Lispro: Participant-specific doses of LY2605541 were administered SC once daily at bedtime for 26 weeks.
  Participant-specific doses of Insulin Lispro were administered SC for preprandial and supplemental doses for 26 weeks.
- Insulin Glargine + Insulin Lispro: Participant-specific doses of Insulin Glargine were administered SC once daily at bedtime for 26 weeks.
  Participant-specific doses of Insulin Lispro were administered SC for preprandial and supplemental doses for 26 weeks.
Arm/Group | LY2605541 + Insulin Lispro | Insulin Glargine + Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 79/691 | 63/677
Other Adverse Events (participants affected / at risk) | 408/691 | 406/677
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2605541 + Insulin Lispro (N=691) | Insulin Glargine + Insulin Lispro (N=677)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (4) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Panophthalmitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bezoar (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (2)
Cellulitis (Infections and infestations) | 3 (6) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 18 (21) | 12 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/315 (1) | 0/273 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/376 (1) | 0/404 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/376 (0) | 1/404 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (4) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/315 (0) | 1/273 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 + Insulin Lispro (N=691) | Insulin Glargine + Insulin Lispro (N=677)
Diabetic retinopathy (Eye disorders) | 7 (8) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 9 (9) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 24 (27) | 19 (22)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 16 (16) | 9 (10)
Vomiting (Gastrointestinal disorders) | 11 (11) | 10 (13)
Asthenia (General disorders) | 0 (0) | 7 (7)
Fatigue (General disorders) | 6 (8) | 16 (16)
Oedema peripheral (General disorders) | 11 (11) | 26 (31)
Pyrexia (General disorders) | 8 (8) | 7 (7)
Bronchitis (Infections and infestations) | 20 (21) | 20 (22)
Gastroenteritis (Infections and infestations) | 8 (9) | 16 (16)
Gastroenteritis viral (Infections and infestations) | 12 (12) | 6 (6)
Influenza (Infections and infestations) | 18 (19) | 16 (17)
Nasopharyngitis (Infections and infestations) | 49 (58) | 63 (69)
Pharyngitis (Infections and infestations) | 3 (3) | 7 (7)
Sinusitis (Infections and infestations) | 16 (19) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 29 (33) | 32 (39)
Urinary tract infection (Infections and infestations) | 18 (19) | 23 (26)
Contusion (Injury, poisoning and procedural complications) | 4 (6) | 8 (9)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 7 (9)
Alanine aminotransferase increased (Investigations) | 11 (12) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 9 (9)
Weight increased (Investigations) | 5 (5) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (17) | 15 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (25) | 23 (25)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 14 (14)
Carpal tunnel syndrome (Nervous system disorders) | 10 (11) | 1 (1)
Dizziness (Nervous system disorders) | 9 (11) | 10 (10)
Headache (Nervous system disorders) | 12 (12) | 19 (20)
Hypoaesthesia (Nervous system disorders) | 7 (8) | 7 (9)
Depression (Psychiatric disorders) | 4 (4) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 9 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (8)
Hypertension (Vascular disorders) | 14 (16) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days